CLINICAL TRIAL: NCT06100926
Title: Effectiveness of Virtual Reality (VR) in Non-oncologic Chronic Musculoskeletal Pain: a Randomized Controlled Trial in Fibromyalgia
Brief Title: Effectiveness of Virtual Reality (VR) in Non-oncologic Chronic Musculoskeletal Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Collaborators: University of Udine (Other)
Responsible Party: Principal Investigator, Luca Quartuccio, Deputy Director of the Rheumatology Division, Azienda Sanitaria-Universitaria Integrata di Udine
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 131/2023
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Musculoskeletal Pain; Fibromyalgia, Primary
MeSH Terms: conditions — Musculoskeletal Pain; Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Active Comparator): subjects who undergo virtual reality immersion scene ab initio
  Interventions: Device: software
- control group (Other): subjects who undergo virtual reality immersion scene in a second phase
  Interventions: Device: software

INTERVENTIONS:
Device: software — virtual reality scene

SUMMARY:
Treatment options for chronic non-oncologic musculoskeletal pain are varied and include both pharmacological and non-pharmacological interventions, such as physical activity and psychotherapy. In clinical practice, the prevalent approach is pharmacological, based mainly on the use of pain modulators, such as antidepressants, cannabinoids and anti-epileptics, and on the use of traditional painkillers such as NSAIDs and opioids. In particular, the latter are still widely prescribed in clinical practice. Initially very effective in combating fibromyalgia pain, opioids, when taken chronically, lead to the development of tolerance with the need for the patient to gradually increase the dosage or switch to more powerful active drugs to obtain the same effect. In the face of fleeting and limited benefits, the risk, therefore, is that of falling back into a framework of abuse with consequent negative impact on both health and social status. In this context, the non-pharmacological approach plays a role of primary importance. In particular, exercise is currently recommended as one of the most effective management strategies. However, the implementation of exercise as a treatment for chronic pain is significantly hampered by poor patient compliance. Another non-pharmacological strategy is biofeedback (BF); however, although existing data support the use of BF, in clinical practice the results obtained have not supported expectations. A solution to these limitations could come from virtual reality (VR), an innovative method capable of simulating real-world situations and cognitive and motor tasks in a safe and stimulating environment, making the completion of activities rewarding and benefiting all those patients who need motor rehabilitation or musculoskeletal pain management.

This is a single-center interventional randomized device-controlled study, with two study arms:

* The treatment group: subjected to 5 days of VR experience and subsequently monitored using questionnaires until the 15th day after the end of the experience.
* The control group: initially placed on hold and subsequently also subjected to 5 days of VR experience only when the treatment group has finished its shift; subsequently each patient will be monitored until the 15th day after the end of the experience.

Primary endpoint:

- Demonstration of a pain change of at least 30% according to the VAS scale (0-100) in patients undergoing VR compared to those not undergoing VR.

Inclusion criteria - Patients aged 18-50 years who complain of chronic musculoskeletal pain lasting at least three months, without diagnosis of inflammatory causes Exclusion criteria

* Concomitant diagnosis of major psychiatric pathologies with the exception of anxiety-depressive disorder;
* Concomitant diagnosis of neurological pathologies;
* Concomitant diagnosis of inflammatory rheumatological diseases that may cause chronic pain.

Statistical analysis On the basis of the primary endpoints set, it is planned to enroll a sample of 20 patients, 10 per treatment group, considering an alpha error of 0.05 and a power of 80%. Considering a dropout of approximately 2 patients, a final sample of 24 patients is considered, 12 for each group.

Comparisons between the two groups of patients will be performed using parametric or non-parametric statistical tests, based on the distribution of the variables, using the Student or Mann-Whitney t test for continuous variables, and Chi-square or Fischer, for variable dichotomous or ordinal. Any correlations will be determined through the calculation of the Odds Ratio.

ELIGIBILITY:
Inclusion Criteria:

Volunteers aged between 18-50 years who suffer from non-cancer musculoskeletal chronic pain and meet the 2016 Modified ACR Diagnostic Criteria for Fibromyalgia will be included in the analysis.

Exclusion Criteria:

* Concomitant diagnosis of major psychiatric disorders except for anxiety-depressive disorder;
* Concomitant diagnosis of neurological disorders;
* Concomitant diagnosis of inflammatory rheumatologic diseases that may cause chronic pain;
* Concomitant diagnosis of severe heart diseases;
* Concomitant diagnosis of epilepsy;
* Concomitant diagnosis of issues related to reality perception;
* Substance addiction

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain change | 0-20 days
  Pain change of at least 30% according to the VAS scale (0-100) in subjects undergoing VR compared to those not undergoing VR.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Division, Udine, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: Yes
The individual, de-identified patient data supporting the findings presented in this article will be accessible to researchers whose intended use of the data has received approval from the corresponding author, along with a signed data access agreement. Access will be granted exclusively for the purposes specified in the approved proposal. For inquiries or to submit proposals, please contact the corresponding author directly.
Supporting Information: Study Protocol, SAP, CSR